CLINICAL TRIAL: NCT00221182
Title: Phase I / II Clinical Trial Regarding Vascular Regeneration Therapy by Transplantation of Autologous Peripheral Blood Endothelial Progenitor Cells (CD34+ Cells) in No-Option Patients With Chronic Myocardial Ischemia
Brief Title: Stem Cell Study for Patients With Heart Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow recruitment of the study subjects
Sponsor: Foundation for Biomedical Research and Innovation (Other)
Collaborators: Institute of Biomedical Research and Innovation, Kobe, Hyogo, Japan (Other); Kobe City General Hospital (Other); Okayama University School of Medicine (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI CAD 04-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Chest Pain; Chronic Myocardial Ischemia; Coronary Artery Disease; Angina; Myocardial Infarction
Keywords: Angina; Heart diseases; Pain; Vascular diseases
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Angina Pectoris; Myocardial Infarction; Heart Diseases; Pain; Vascular Diseases

INTERVENTIONS:
Genetic: Autologous peripheral blood CD34 positive cell therapy

SUMMARY:
The purpose of this study is to determine if stem cell therapy with your own cells (autologous cells) delivered with a catheter to regions of the heart with poor blood flow will be safe and if it will relieve your chest pain, increase the blood flow, and/or improve the cardiac contractility (function) by regenerating blood vessels in your heart.

DETAILED DESCRIPTION:
Chronic myocardial ischemia (MI) is a progressive disease, which arises as a result of atherosclerosis in coronary arteries. Prognosis of chronic MI is poor, and no effective treatments have been established in patients who are not eligible for the traditional revascularization therapies such as angioplasty and bypass procedures due to the inappropriate anatomy of the coronary arteries or frequent reocclusion following revascularization. Therefore, it is necessary to establish novel revascularization treatment to improve prognosis of the no-option patients. We will study the safety and clinical efficiency of vascular regeneration by means of transplantation of autologous peripheral blood endothelial progenitor cells (CD34 positive cells) in patients with severe chronic coronary artery disease (CAD) who are not eligible for traditional revascularization treatments. The primary endpoint is the severity of myocardial ischemia identified by sestamibi SPECT stress myocardial scintigraphy and the evaluation of adverse effect rates, while the secondary endpoints are evaluation of CCSAS and NYHA classification, regional myocardial blood flow as revealed by PET scan, and various left ventricular function indices.

ELIGIBILITY:
Inclusion Criteria:

-Chronic severe CAD patients fulfilling all the following criteria are considered suitable for inclusion in the study.

1. At least 6 months since last episode of myocardial infarction or at least 3 months since initial anginal episode.
2. Patients fulfilling either of the following criteria based on the extent of CAD by coronary angiography and LVEF by echocardiography.

   * Patients with single vessel CAD and LVEF < 50%
   * Patients with multivessel CAD
3. Reversible myocardial ischemia as revealed by sestamibi SPECT stress myocardial scintigraphy.
4. Patients for whom angioplasty and bypass are not indicated because of anatomical or procedural reasons or frequent reocclusion/restenosis following traditional revascularization.
5. Age is between 20 and 80 (at time of consent).
6. Exercise tolerance time (ETT) duration ≥ 3 minutes and < 13 minutes on a modified Bruce protocol on 2 consecutive tests (> 24 hours but < 2 weeks apart), with the difference between the 2 exercise times within 25% of their mean (Patients should not be informed of exercise restrictions required for entry into the study).
7. Patients who can give informed consent themselves in writing.

Exclusion Criteria:

* Any one of the following exclusion criteria is sufficient to disqualify a patient from the study.

  1. Sustained ventricular tachycardia in a 24-hour ECG.
  2. Chronic atrial fibrillation.
  3. Less than 6 months since last episode of cerebral infarction.
  4. Less than 6 months since last coronary angioplasty or less than 3 months since last bypass surgery.
  5. Patients with unstable angina, with a treatment rating of 3 in the Braunwald system (refer to 5.4.), but a severity of III and a clinical rating of B or C.
  6. Presence of left ventricular thrombus by echocardiography
  7. Patients with a malignant tumor*.
  8. Patients with diabetic proliferating retinopathy** (new Fukuda classification BI to BV).
  9. Patients with chronic rheumatoid arthritis.
  10. Patients with a history of severe allergic reactions or side effects to G-CSF preparations or apheresis.
  11. Patients with hematological disease (leukemia, myeloproliferative disease, or myelodysplastic syndromes).
  12. Patients currently suffering from or having a history of interstitial pneumonitis.
  13. Patients for whom cranial MRA reveals cerebral aneurysm.
  14. Patients for whom abdominal CT or ultrasonography reveals splenomegaly.
  15. Patients with cirrhosis of the liver.
  16. Patients who cannot discontinue Warfarin.
  17. Leukocytes less than 4,000/µL or exceeding 10,000/µL.
  18. Platelets less than 100,000/µL.
  19. Hemoglobin less than 10 g/dL.
  20. AST (GOT) exceeding 100 IU/L or ALT (GPT) exceeding 100 IU/L.
  21. Patients for whom it is impossible to perform both cardiac MRI and left ventriculography (LVG) (see 9.2.4 for cardiac MRI details and 9.2.9 for LVG details).
  22. Patients with gate disturbance for reasons other than CAD (such as critical limb ischemia, sciatic neuralgia, or vasculitis), making exercise tolerance evaluation on a treadmill with stress ECG difficult.
  23. Pregnant or nursing patients, those who may be pregnant, or those who plan on becoming pregnant before the end of the study period.
  24. Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Efficacy: Severity of myocardial perfusion abnormality by sestamibi SPECT stress myocardial scintigraphy
Safety: Severe adverse events within 4 weeks after cell therapy

SECONDARY OUTCOMES:
CCSAS (Canada Cardiovascular Society Anginal Score)
NYHA (New York Heart Association) classification
Exercise tolerance by treadmill
Left ventricular function by cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Asahara, M.D., Principal Investigator — Foundation for Biomedical Research and Innovation
Locations (3):
- Japan (3):
  - Kobe Institute of Biomedical Research and Innovation, Kobe, Hyogo-Pref.
  - Kobe City General Hospital, Kobe, Hyōgo
  - Okayama University School of Medicine, Okayama, Okayama-ken

REFERENCES:
- [Background] Asahara T, Kawamoto A. Endothelial progenitor cells for postnatal vasculogenesis. Am J Physiol Cell Physiol. 2004 Sep;287(3):C572-9. doi: 10.1152/ajpcell.00330.2003. PMID 15308462
- [Background] Kawamoto A, Tkebuchava T, Yamaguchi J, Nishimura H, Yoon YS, Milliken C, Uchida S, Masuo O, Iwaguro H, Ma H, Hanley A, Silver M, Kearney M, Losordo DW, Isner JM, Asahara T. Intramyocardial transplantation of autologous endothelial progenitor cells for therapeutic neovascularization of myocardial ischemia. Circulation. 2003 Jan 28;107(3):461-8. doi: 10.1161/01.cir.0000046450.89986.50. PMID 12551872
- [Background] Kawamoto A, Gwon HC, Iwaguro H, Yamaguchi JI, Uchida S, Masuda H, Silver M, Ma H, Kearney M, Isner JM, Asahara T. Therapeutic potential of ex vivo expanded endothelial progenitor cells for myocardial ischemia. Circulation. 2001 Feb 6;103(5):634-7. doi: 10.1161/01.cir.103.5.634. PMID 11156872
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398